CLINICAL TRIAL: NCT05414890
Title: Comparison of the Specificity, Sensitivity, and Clinical Correlation of Cell-based Assay (CBA) and CBA-TSA (Tyramide Signal Amplification) in Detecting AQP4, MOG, and NMDAR-IgG in Central Nervous System Diseases; a National Multicenter Study
Brief Title: Sensitivity and Specificity of TSA-CBA for Autoantibodies Against Neural Antigen Determination
Acronym: STAND
Status: Unknown | Type: Observational
Last Known Status: Recruiting
Sponsor: Beijing Tiantan Hospital (Other)
Collaborators: Tianjin Medical University General Hospital (Other)
Responsible Party: Sponsor
Other Study IDs: IRB2022-YX-066-01
Record Dates: First submitted 2022-05-31; First posted 2022-06-10 (Actual); Last update posted 2022-06-10 (Actual); Status verified 2022-06

CONDITIONS: NMO Spectrum Disorder; NMDA-R Encephalitis; Diagnostic Self Evaluation; Immune System Diseases; Nervous System Diseases; Autoimmune Diseases of the Nervous System; Autoimmune Diseases
MeSH Terms: conditions — Neuromyelitis Optica; Immune System Diseases; Nervous System Diseases; Autoimmune Diseases of the Nervous System; Autoimmune Diseases

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (2):
- Cell Based Assay (CBA): The sera samples from patients and control subjects, upon clinic visits, as well as during follow up, will be randomly numbered. All samples will be blindly tested with CBA by different operators.
- CBA-TSA Assay: The sera samples from patients and control subjects, upon clinic visits, as well as during follow up, will be randomly numbered. All samples will be blindly tested with CBA-TSA by different operators.
  Interventions: Diagnostic Test: CBA-TSA

INTERVENTIONS:
Diagnostic Test: CBA-TSA — Compare the specificity, sensitivity, and clinical correlation between CBA and CBA-TSA, in detecting AQP4, MOG, and NMDAR IgG
  Groups: CBA-TSA Assay

SUMMARY:
Determination of autoantibodies against fragments derived from neurons, glia, and myelin sheath is instrumental in aiding diagnosis, differential diagnosis, as well as determining disease status of neuromyelitis optica spectrum disorders (NMOSD), myelin oligodendrocyte glycoprotein antibody-associated disease (MOGAD), autoimmune encephalitis (AE). Cell based assay (CBA) has been frequently recommended to detect autoantibodies of neuroantigens in the aforementioned neurological disorders. However, antibodies with low abundance or low affinity often fall beyond the threshold of CBA and pose significant challenges in practice. To this end, the investigators adopted a tyramide signal amplification (TSA) technology with the basis of CBA to improve sensitivity. The preliminary results suggest that this TSA-CBA platform is superior to conventional CBA in registered signals of the titer autoantibodies. In elevating the sensitivity, TSA-CBA also preserves antigen confirmation. This prospective study is launched to compare the sensitivity, specificity, clinical correlation between CBA and CBA-TSA, in determining autoantibodies against aquaporin 4 (AQP4-IgG), myelin oligodendrocyte glycoprotein (MOG-IgG), N-methyl-D-aspartate receptor (NMDAR-IgG) in a multicenter, double-blind setting.

DETAILED DESCRIPTION:
Participants: The sera of patients with CNS demyelinating autoimmune diseases (NMOSD, MOGAD, AE).

Primary aim: 1) Compare the specificity, sensitivity, and clinical correlation between CBA and CBA-TSA, in detecting AQP4, MOG, and NMDAR IgG. 2) Analyze the advantage of CBA-TSA assay over conventional CBA in detecting antibodies to AQP4, MOG, and NMDAR IgG with low abundance and low affinity.

Secondary aim: Comparison of the turn-around time and the cost of CBA and CBA-TSA in detecting AQP4, MOG, and NMDAR IgG.

Study design: Multicenter, double-blind, CBA and CBA-TSA methodology comparison

Total cases:

1. 1000 patients with suspected NMOSD, MOGAD and 1000 patients with suspected autoimmune encephalitis (AE) will be recruited.
2. 500 normal subjects will be recruited.

Trial Period: The trial recruiting duration is 1-2 years.

Research reagents: 1. The reagents for of AQP4, MOG or NMDAR IgG antibody detection via CBA have been developed and validated by the joint effort of Bejing Tiantan Hospital, Tianjin General Hospital, and Tianjin New Terrain Biological Technology Co., Ltd, China , will be adopted by this study. 2. The CBA-TSA antibody IgG assay developed by the three entities and will be adopted for this study

Groups: The sera samples from patients and control subjects, upon clinic visits, as well as during follow up, will be randomly numbered. All samples will be blindly tested with CBA-TSA and CBA by different operators.

Study Steps:

1. Patients recruiting: 1000 patients with suspected NMOSD, MOGAD and 1000 patients with suspected AE will be recruited according to inclusion/exclusion criteria.
2. CBA/CBA-TSA assay: Sera samples from patients and control subjects will be randomly numbered and divided into 3 equal parts (500 ul/part). All samples will be tested with CBA-TSA and CBA by different blinded operators; original value, control value, turn-around time and cost will all be recorded. The difference comparison between CBA and CBA-TSA was completed by Bejing Tiantan Hospital.
3. Statistical Methods: Each center will provide feedback of the clinical diagnosis and treatment data of the participants to the investigator. The investigator will complete the evaluation of respective clinical correlation of the CBA and CBA-TSA methods. The statistics and operation of the project are supervised by a third-party audit company.

ELIGIBILITY:
Inclusion Criteria:

1. The patients with suspected NMOSD, MOGAD and AE will be recruited.
2. Male and female patients, ≥ 18 years old.

Exclusion Criteria:

1. Abnormal sera, such as hemolysis or lipemia, which will affect the final interpretation of CBA and CBA-TSA;
2. The samples with incomplete clinical data that would affect the disease characterization.

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Study Population: The patients with CNS demyelinating autoimmune diseases (NMOSD, MOGAD, AE)
Sampling Method: Probability Sample
Enrollment: 2500 (Estimated)
Dates: Start 2022-06-30 (Estimated); Primary Completion 2024-01-30 (Estimated); Study Completion 2024-06-30 (Estimated)

PRIMARY OUTCOMES:
CBA-TSA is consistent with CBA in terms of specificity and clinical correlation in detecting autoantibodies. | 2022.6.30-2024.6.30
  Comparsion the specificity, sensitivity, positive likelihood ratio (LR), negative LR and clinical correlation of CBA and CBA-TSA assay in autoantibodies detection of AQP4, MOG, NMDAR respectively.
CBA-TSA is superior to CBA for detecting antibodies to AQP4, MOG, and NMDAR IgG with low abundance and low affinity. | 2022.6.30-2024.6.30
  Comparsion the sensitivity of CBA and CBA-TSA assay in detecting the AQP4, MOG or NMDAR IgG in low abundance and low affinity.

SECONDARY OUTCOMES:
Compared with CBA, CBA-TSA uses a smaller sample and costs less, but the experiment turn-around time takes longer. | 2022.6.30-2024.6.30
  Comparsion the detection time, costs and sample usage of CBA and CBA-TSA assay in autoantibodies detection of AQP4, MOG, NMDAR.

CONTACTS AND LOCATIONS:
Locations (1):
- Beijing Tiantan Hospital, Beijing, Beijing Municipality, China

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Zhang C, Tian DC, Yang CS, Han B, Wang J, Yang L, Shi FD. Safety and Efficacy of Bortezomib in Patients With Highly Relapsing Neuromyelitis Optica Spectrum Disorder. JAMA Neurol. 2017 Aug 1;74(8):1010-1012. doi: 10.1001/jamaneurol.2017.1336. PMID 28692708
- [Background] Zhang C, Zhang M, Qiu W, Ma H, Zhang X, Zhu Z, Yang CS, Jia D, Zhang TX, Yuan M, Feng Y, Yang L, Lu W, Yu C, Bennett JL, Shi FD; TANGO Study Investigators. Safety and efficacy of tocilizumab versus azathioprine in highly relapsing neuromyelitis optica spectrum disorder (TANGO): an open-label, multicentre, randomised, phase 2 trial. Lancet Neurol. 2020 May;19(5):391-401. doi: 10.1016/S1474-4422(20)30070-3. PMID 32333897